CLINICAL TRIAL: NCT04330196
Title: Deciphering the Enigma of Postprandial Hyperinsulinaemic Hypoglycaemia After Bariatric Surgery, Part 1 C: Effect of Postprandial Hypoglycaemia on Driving Performance.
Brief Title: Effect of Postprandial Hyperinsulinaemic Hypoglycaemia on Driving Performance.
Acronym: DEEP1C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lia Bally (Other)
Responsible Party: Sponsor-Investigator, Lia Bally, Professor, Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: DEEP1C
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Roux-en-Y Gastric Bypass; Postprandial Hypoglycemia; Driving Impaired
MeSH Terms: conditions — Hypoglycemia | interventions — Glucose Tolerance Test

STUDY DESIGN:
Intervention Model Description: Participants will undergo two experiments in random order. In the experiments, driving performance will be assessed after administration of glucose (intervention arm) or aspartame (control arm).
Who Masked: Participant
Masking Description: Participants will be masked to the type of beverage ingested at each visit (200ml of water containing glucose or aspartame). Furthermore, participants will be masked to glucose levels throughout the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucose condition (Experimental): In the experimental condition patients ingest 200ml of water containing 75g of glucose
  Interventions: Diagnostic Test: Oral glucose tolerance test
- Control condition (Placebo Comparator): In the control condition patients ingest 200ml of water sweetened with 700mg of aspartame
  Interventions: Diagnostic Test: Ingestion of placebo

INTERVENTIONS:
Diagnostic Test: Oral glucose tolerance test — Participant ingests 75g of glucose
  Arms: Glucose condition
Diagnostic Test: Ingestion of placebo — Participant ingests 700mg of aspartame
  Arms: Control condition

SUMMARY:
The primary objective of this study is to assess the effect of the natural course of postprandial hypoglycemia vs. a postprandial euglycaemic condition on driving performance in individuals with confirmed postprandial hyperinsulinaemic hypoglycaemia after gastric-bypass surgery.

DETAILED DESCRIPTION:
Despite the increasing prevalence of postprandial hyperinsulinaemic hypoglycaemia (PHH), clinical implications are still unclear. Anecdotal evidence from patients with PHH suggest a high burden for these patients due to the recurrent hypoglycaemias with possibly debilitating consequences. It is well established, that even mild hypoglycaemia (plasma glucose of 3.4mmol/l) in diabetic and non-diabetic significantly impairs cognitive-motor functioning. Of note, some of the cognitive aspects remain impaired for up to 75min, even when the hypoglycaemia is corrected. In addition to the hypoglycaemic blood glucose levels per se, the dynamics of the hypoglycaemia occurrence appears to play a role. It was shown in individuals with type 1 diabetes, that cognitive functions are affected more during a fast-fall than slow fall hypoglycaemia in the postprandial state.

Driving is a frequent daily activity which integrates various mental function including visual and auditory processing, motor skills, reasoning and problem solving. Due to the potentially dangerous consequences, avoidance of hypoglycaemia-induced driving mishaps is of uttermost importance. Several studies have evaluated the impact of induced, controlled hypoglycaemia in individuals with type 1 diabetes on driving performance using driving simulators but data in PHH patients are currently lacking. Assessing the potential impact of the natural course of postprandial hypoglycaemia on driving performance in PHH patients will contribute to a better understanding of the consequences and relevance of this problem. The investigator will test the hypothesis whether driving performance during the postprandial glucose dynamics is impaired in patients with confirmed PHH.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Roux-en-Y gastric bypass ≥1 year ago
* PHH defined as postprandial plasma or sensor glucose<3.0mmol/l according to the International Hypoglycaemia Study Group (1) and exclusion of other causes of hypoglycaemia
* Possession of a valid Swiss driver's license. Passed driver's examination at least 3 years before study inclusion. Active driving in the last 6 months before the study.

Exclusion Criteria:

* Clinically relevant weight changes (≥5%) within the past 3 months
* Incapacity to give informant consent
* Historical or current diabetes based on HbA1c ≥6.5% without glucose-lowering treatment
* Haemoglobin level below 11 g/dl
* Ongoing treatment with glucose-lowering drugs, anorectic drugs, steroids or any medications known to affect gastric motility
* Active heart, lung, liver, gastrointestinal, renal or neurological disease
* Inability to follow study procedures
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
Estimated difference in driving performance across driving features over the glycemic trajectory after glucose vs. aspartame intake | From -15 to 150 minutes after glucose/aspartame intake
  The pooled effect (z-score difference), which is the compound change in driving performance across driving features between the glucose and aspartame condition, will be calculated using a Bayesian hierarchical regression model

SECONDARY OUTCOMES:
Hypoglycemic symptoms over the glycemic trajectory after glucose vs. aspartame intake | From -15 to 180 minutes after glucose/aspartame intake
  Hypoglycemic symptoms will be rated using the Edinburgh Hypoglycemia Symptom Scale (minimum score=11, maximum score=77, a higher score, means more symptoms)
Cognitive test performance after glucose vs. aspartame intake | 135 minutes after glucose/aspartame intake
  Cognitive function will be assessed using the Digit Symbol Substitution Test

OTHER OUTCOMES:
Time course of the hormonal response after glucose/aspartame intake | From -15 to 120 minutes after glucose/aspartame intake
  Insulin, C-peptide, Adrenalin, Noradrenalin, Glucagon, Cortisol, Growth hormone, PYY will be measured in pre-defined timepoints
Heart rate after glucose/aspartame intake | From -15 to 180 minutes after glucose/aspartame intake
  An ECG will be used to measure heart rate after glucose and aspartame intake

CONTACTS AND LOCATIONS:
Overall Officials: Lia Bally, MD, PhD, Principal Investigator — University Hopsital Bern, University of Bern
Locations (1):
- Department of Diabetes, Endocrinology, Clinical Nutrition and Metabolism, Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No